CLINICAL TRIAL: NCT05149495
Title: Maintenance of Remission After Discontinuation of Somatostatin Analogues in the Treatment of Relapsing GH Pituitary Adenomas After Surgery
Brief Title: Somatostatin Analogues in the Treatment of Relapsing GH Pituitary Adenomas After Surgery
Acronym: STOP-SST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8409
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Acromegaly
Keywords: Acromegaly; Pituitary microadenoma; Pituitary macroadenoma; Somatostatin analogues; Hormonal control
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At present there are no recommendations regarding the possibility of discontinuing treatment in cases of recurrent acromegaly with good hormonal control. Discontinuation of treatment is therefore most often decided by the practitioner, on the basis of his experience and knowledge of the patient, the long-term course with somatostatin analogues being very little described.

Thus, although hormonal control is achieved in a majority of cases under medical treatment, we do not know if it is possible to stop treatment and in this case how the pathology evolves. It would appear that approximately 40% of patients defined as very good responders to somatostatin analogues may gradually space their injections.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Having been seen at least once in consultation in the Internal Medicine, Endocrinology and Nutrition department of Hautepierre Hospital
* Subject operated for a pituitary adenoma at the HUS between 01/01/2000 to 09/01/2021
* In whom biological confirmation of recurrence has been demonstrated
* Patient not having expressed his opposition, after information, to the reuse of his data for scientific research purposes.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Treatment pre and / or post surgery by radiotherapy
* No recurrence
* No treatment with a somatostatin analogue for recurrence
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject operated for a pituitary adenoma at the HUS between 01/01/2000 to 09/01/2021
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Study of the clinical and biological evolution, after discontinuation of treatment with somatostatin analogues, of acromegalic patients with recurrence after surgery. | Files analysed retrospectively from January 01, 2000 to September 01, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BALTZINGER, MD, Principal Investigator — Service Médecine Interne, Endocrinologie et Nutrition - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service Médecine Interne, Endocrinologie et Nutrition - Hôpitaux Universitaires de Strasbourg, Strasbourg, France